CLINICAL TRIAL: NCT06369207
Title: Evaluation of Reflux Transmission Pathways in Chronic Venous Insufficiency Patients Secondary to Saphenofemoral Reflux, Presenting to Vascular Surgery Clinics of Golestan Province From 2022 Till 2023
Brief Title: Investigation of the Transmission Pathways of Reflux in Patients With Chronic Venous Insufficiency
Status: Completed | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Pezhman Kharazm, MD, Vascular Surgeon, Golestan University of Medical sciences
Other Study IDs: 113454
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Venous Insufficiency
Keywords: venous insufficiency; reflux; ultrasonographic mapping; saphenofemoral junction
MeSH Terms: conditions — Venous Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic venous insufficiency (CVI) is one of the most common medical problems in adults that occurs secondary to the reflux of blood through incompetent valves of lower extremity veins. The most common involved valve is the valve located at the saphenofemoral junction. Although the pathway of reflux transmission is not the same in all patients, the removal or ablation of the greater saphenous vein (GSV) is considered a standard treatment in these patients. However, in patients whose reflux is transmitted to branches other than GSV, this treatment leads to the unnecessary destruction of a competent segment of GSV in addition to remaining at least some segments of incompetent veins. So, in this study, the investigators intend to investigate the different pathways of reflux transmission in chronic venous insufficiency patients who are candidates for GSV ablation/stripping because of saphenofemoral junction insufficiency. This cross-sectional study will be conducted with a descriptive-analytical approach. .

DETAILED DESCRIPTION:
Chronic venous insufficiency is one of the most common medical diseases in adults, which severely affects the quality of life of affected patients. What causes symptoms in this disease is the reflux of blood through incompetent valves located in the lower extremity veins. The most common cause is saphenofemoral valve insufficiency.

Although the pathway of reflux transmission is not the same in all patients, the removal of the greater saphenous vein (GSV) is considered a standard treatment according to the guidelines. This treatment leads to unnecessary destruction of the great saphenous vein and failure to correct the pathology in patients whose reflux exited the GSV along its transmission pathway. According to this issue, in this study, the investigators intend to investigate the different pathways of reflux transmission in chronic venous insufficiency patients who are candidates for GSV ablation/stripping because of saphenofemoral junction insufficiency according to the ultrasonographic exam. This cross-sectional study will be conducted with a descriptive-analytical approach on approximately 50 participants. Before surgery, patients are subjected to ultrasonographic mapping to check the pathway of reflux transmission and their related information is recorded. Other demographic information will also be recorded in the relevant checklist. Finally, the data will be analyzed in SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Age>18.
* Chronic Venous Insufficiency with a clinical grade of 3 (varicosity) or more.
* Documentation of saphenofemoral junction insufficiency on Doppler ultrasound performed by a radiologist.
* Patient consent.

Exclusion Criteria:

- History of DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included participants are visited the day before surgery and venous mapping is performed for the patient by the vascular surgeon. The reflux pathway is marked on the skin and information regarding the anatomic characteristics of the reflux are recorded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Determination of reflux transmission pathways in CVI patients with SFJ incompetency | one year
  Determining the transmission pathways of reflux in patients with chronic venous insufficiency secondary to saphenofemoral reflux referring to vascular surgery clinics in Golestan province from 2022 to 2023

SECONDARY OUTCOMES:
Anatomic variations of GSV in CVI patients with SFJ incompetency | one year
  Determining the frequency of anatomical variations of the great saphenous vein in patients with chronic venous insufficiency secondary to saphenofemoral reflux
Prevalence of reflux along GSV main trunk in CVI patients with SFJ incompetency | one year
  Determining the frequency of reflux in the main trunk of the great saphenous vein in patients with chronic venous insufficiency secondary to saphenofemoral reflux.
Prevalence of reflux along accessory saphenous veins in CVI patients with SFJ incompetency | one year
  Determining the frequency of reflux along accessory saphenous veins in patients with chronic venous insufficiency secondary to saphenofemoral reflux.

CONTACTS AND LOCATIONS:
Locations (1):
- Pezhman Kharazm, MD, Gorgan, Golestan Province, Iran